CLINICAL TRIAL: NCT04949191
Title: An Open-Label, Multicenter, Rollover Study to Provide Continued Treatment for Participants With Advanced Malignancies Previously Enrolled in Studies of Pemigatinib
Brief Title: The Purpose of the Study is to Continue to Provide Pemigatinib to Patients With Advanced Malignancies.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A business decision due to availability of commercial drug and other options for accessing study drug treatment.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 54828-801
Record Dates: First submitted 2021-06-25; First posted 2021-07-02 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Advanced Malignancies
Keywords: pemigatinib
MeSH Terms: interventions — pemigatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Study Treatment 1: Pemigatinib (INCB054828) (Experimental): Pemigatinib will be taken orally once daily
  Interventions: Drug: Pemigatinib
- Study Treatment 2: Pemigatininb+ Retifanlimab (Experimental): Participants rolling over from study INCB 54828-101 only will receive pemigatinib once daily and retifanlimab will be administered once every 4 weeks
  Interventions: Drug: Pemigatinib; Drug: Retifanlimab
- Study Treatment 3: Pemigatininb + Pembrolizumab (Experimental): Participants rolling over from study INCB 54828-101 only will receive pemigatinib once daily and pembroluzimab as per dosage instructions.
  Interventions: Drug: Pemigatinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pemigatinib — Pemigatinib tablets taken by mouth once daily as per protocol
  Other Names: INCB054828
Drug: Retifanlimab — Retifanlimab is administered over 60 minutes once every 4 weeks (Day 1 of a 28-day cycle)
  Other Names: INCMGA0012
  Arms: Study Treatment 2: Pemigatininb+ Retifanlimab
Drug: Pembrolizumab — Commercially labeled products
  Arms: Study Treatment 3: Pemigatininb + Pembrolizumab

SUMMARY:
Safety and tolerability of pemigatinib.in monotherapy or combination in patients that have participated in a previous parent study to treat advanced malignancies.

DETAILED DESCRIPTION:
A Phase 2 Open-Label, Multicenter, Rollover Study to evaluate the long term safety and tolerability of Pemigatinib and to provide Continued Treatment for Participants With Advanced Malignancies Previously Enrolled in Studies of Pemigatinib

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled and receiving treatment in an Incyte-sponsored clinical study (parent protocol) of pemigatinib as monotherapy or combination therapy.
* Currently benefiting from and tolerating treatment with pemigatinib, as determined by the investigator.
* Demonstrated compliance, as assessed by the investigator, with the parent protocol requirements.
* Willingness and ability to comply with scheduled visits, treatment plans, and any other study procedures.
* Currently have no evidence of progressive disease, as determined by the investigator, following treatment with pemigatinib as monotherapy or combination therapy.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Able to access pemigatinib commercially or outside of a clinical trial.
* Permanently discontinued from the parent protocol for any reason.
* No longer meet the inclusion/exclusion criteria from the parent protocol if still receiving treatment.
* Women who are pregnant or breastfeeding or participants expecting to conceive or father children within the projected duration of the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Langmuir, Study Director — Incyte Corporation
Locations (10):
- United States (5):
  - John Wayne Cancer Institute, Santa Monica, California
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Md Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - Virginia Cancer Specialists, Pc, Fairfax, Virginia
- The Finsen Centre National Hospital, Copenhagen, Denmark
- Italy (3):
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - Istituto Nazionale Tumori Regina Elena Irccs, Rome
  - Azienda Ospedaliera Universitaria Senese Policlinico Santa Maria Alle Scotte, Siena
- Kanagawa Cancer Center, Yokohama, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were actively receiving treatment with pemigatinib (monotherapy or in combination with pembrolizumab) under a parent protocol, were receiving clinical benefit in those trials, and who did not have access to pemigatinib (as monotherapy or as combination therapy) outside of a clinical trial were enrolled.
Pre-assignment Details: This study was conducted at 9 sites in 4 countries.
Groups:
- Pemigatinib 6 mg Monotherapy: Participants originally enrolled in a parent study (54828-201 [NCT02872714], 54828-202 [NCT02924376], or 54828-207 [NCT03822117]), who received clinical benefit from pemigatinib, and who did not have access to pemigatinib outside of a clinical trial self-administered oral pemigatinib 6 milligrams (mg) once daily (QD), either continuously in 21-day cycles or on a 2-weeks-on therapy/1-week-off therapy schedule in 21-day cycles. Pemigatinib was administered at the same dose received in the parent studies until documented disease progression or unacceptable toxicity.
- Pemigatinib 9 mg Monotherapy: Participants originally enrolled in a parent study (54828-201 [NCT02872714], 54828-202 [NCT02924376], or 54828-207 [NCT03822117]), who received clinical benefit from pemigatinib, and who did not have access to pemigatinib outside of a clinical trial self-administered oral pemigatinib 9 mg QD, either continuously in 21-day cycles or on a 2-weeks-on therapy/1-week-off therapy schedule in 21-day cycles. Pemigatinib was administered at the same dose received in the parent studies until documented disease progression or unacceptable toxicity.
- Pemigatinib 13.5 mg Monotherapy: articipants originally enrolled in a parent study (54828-201 [NCT02872714], 54828-202 [NCT02924376], or 54828-207 [NCT03822117]), who received clinical benefit from pemigatinib, and who did not have access to pemigatinib outside of a clinical trial self-administered oral pemigatinib 13.5 mg QD, either continuously in 21-day cycles or on a 2-weeks-on therapy/1-week-off therapy schedule in 21-day cycles. Pemigatinib was administered at the same dose received in the parent studies until documented disease progression or unacceptable toxicity.
- Pemigatinib Combination: Participants originally enrolled in parent study 54828-101 (NCT02393248), who received clinical benefit from the combination of pemigatinib plus pembrolizumab, and who did not have access to the combination outside of a clinical trial received received the combination of pemigatinib and pembrolizumab. Participants received pembrolizumab intravenously at 200 mg once every 3 weeks on Day 1 of each 21-day cycle. The dose could have been adjusted for toxicity management per commercial labeling. The investigator could have interrupted, modified, or discontinued pembrolizumab with medical monitor approval. Participants self-administered oral pemigatinib 13.5 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. It was permissible to continue pemigatinib administration during the toxicity break of pembrolizumab.
Period: Overall Study
Arm/Group | Pemigatinib 6 mg Monotherapy | Pemigatinib 9 mg Monotherapy | Pemigatinib 13.5 mg Monotherapy | Pemigatinib Combination
Started | 2 | 5 | 2 | 1
Completed | 1 | 3 | 1 | 0
Not Completed | 1 | 2 | 1 | 1
Not completed — Non-compliance with Study Drug | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 1 | 0 | 0
Not completed — Transitioned to Commercial Pemigatinib | 0 | 1 | 0 | 0
Not completed — Sponsor Terminated Study | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The 6 mg (n=2) and 13.5 mg (n=2) monotherapy groups have been combined into a single arm retain participant privacy and reduce the risk of participant re-identification.
Groups:
- Pemigatinib 6 mg and 13.5 mg Monotherapy: Participants originally enrolled in a parent study (54828-201 [NCT02872714], 54828-202 [NCT02924376], or 54828-207 [NCT03822117]), who received clinical benefit from pemigatinib, and who did not have access to pemigatinib outside of a clinical trial self-administered oral pemigatinib 6 milligrams (mg) or 13.5 mg once daily (QD), either continuously in 21-day cycles or on a 2-weeks-on therapy/1-week-off therapy schedule in 21-day cycles. Pemigatinib was administered at the same dose received in the parent studies until documented disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Pemigatinib 6 mg and 13.5 mg Monotherapy | Pemigatinib 9 mg Monotherapy | Pemigatinib Combination | Total
Number analyzed (Participants) | 4 | 5 | 1 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (17.20) | 61.2 (6.30) | NA (NA) — Mean age (SD) cannot be reported for a single participant due to privacy concerns/risk of participant identification. | NA (NA) — Mean (SD) age for the total arm cannot be reported due to privacy concerns/risk of participant identification. The age of the 1 participant in the combination arm could be calculated if the mean (SD) age for the total group and the mean (SD) ages for the participants in the monotherapy arms are known.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | NA — Sex cannot be reported for a single participant due to privacy concerns/risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | 2 | 3 | NA — Sex cannot be reported for a single participant due to privacy concerns/risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | NA — Ethnicity cannot be reported for a single participant due to privacy concerns/risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Not Hispanic or Latino | 4 | 5 | NA — Ethnicity cannot be reported for a single participant due to privacy concerns/risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 0 | 0 | NA — Ethnicity cannot be reported for a single participant due to privacy concerns/risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 2 | 4 | NA — Gender cannot be reported for a single participant due to privacy concerns/risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | 1 | 1 | NA — Gender cannot be reported for a single participant due to privacy concerns/risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black/African-American | 1 | 0 | NA — Gender cannot be reported for a single participant due to privacy concerns/risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. TEAEs were defined as AEs either reported for the first time or the worsening of pre-existing events after the first dose of study drug and until 30 days after the last dose of study drug.
Time Frame: up to at least 30 days after the last dose of study treatment or until toxicities resolve, return to baseline, or are deemed irreversible, whichever was longer (up to 1010 days)
Population: Safety Population: all participants who received at least 1 dose of study treatment in this study
Measure: Count of Participants; unit: Participants
Groups:
- Pemigatinib 13.5 mg Monotherapy: Participants originally enrolled in a parent study (54828-201 [NCT02872714], 54828-202 [NCT02924376], or 54828-207 [NCT03822117]), who received clinical benefit from pemigatinib, and who did not have access to pemigatinib outside of a clinical trial self-administered oral pemigatinib 13.5 mg QD, either continuously in 21-day cycles or on a 2-weeks-on therapy/1-week-off therapy schedule in 21-day cycles. Pemigatinib was administered at the same dose received in the parent studies until documented disease progression or unacceptable toxicity.
Arm/Group | Pemigatinib 6 mg Monotherapy | Pemigatinib 9 mg Monotherapy | Pemigatinib 13.5 mg Monotherapy | Pemigatinib Combination
Number analyzed (Participants) | 2 | 5 | 2 | 1
Participants | 1 | 5 | 1 | 1

ADVERSE EVENTS:
Time Frame: up to 1010 days
Description: Treatment-emergent adverse events (TEAEs), defined as AEs either reported for the first time or the worsening of pre-existing events after the first dose of study drug and until 30 days after the last dose of study drug, have been reported.
Arm/Group | Pemigatinib 6 mg Monotherapy | Pemigatinib 9 mg Monotherapy | Pemigatinib 13.5 mg Monotherapy | Pemigatinib Combination
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/5 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/5 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 5/5 | 1/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemigatinib 6 mg Monotherapy (N=2) | Pemigatinib 9 mg Monotherapy (N=5) | Pemigatinib 13.5 mg Monotherapy (N=2) | Pemigatinib Combination (N=1)
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemigatinib 6 mg Monotherapy (N=2) | Pemigatinib 9 mg Monotherapy (N=5) | Pemigatinib 13.5 mg Monotherapy (N=2) | Pemigatinib Combination (N=1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Corneal erosion (Eye disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Multiple allergies (Immune system disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Nail infection (Infections and infestations) | 0 | 1 | 0 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Porokeratosis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Shoulder fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 4 | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT04949191/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT04949191/SAP_001.pdf